CLINICAL TRIAL: NCT02783547
Title: A Phase 1, Open Label, Multicentre Clinical Trial of SyB C-1101 in Combination With Azacytidine in Patients With Myelodysplastic Syndrome
Brief Title: Combination Therapy of SyB C-1101 and Azacytidine in Patients With Myelodysplastic Syndrome
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was withdrawn due to problems with the manufacture of the investigational drug.
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015001
Record Dates: First submitted 2016-03-06; First posted 2016-05-26 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

ARMS (1):
- SyB C-1101 and Azacytidine (Experimental)
  Interventions: Drug: SyB C-1101 and Azacytidine

INTERVENTIONS:
Drug: SyB C-1101 and Azacytidine — This study is a multi-center open-label study to assess the tolerability of oral administration of SyB C-1101 twice daily from Day 1 to Day 21 in combination with subcutaneous administration or intravenous drip infusion of azacitidine once daily at a dose of 75 mg/m2 (body surface) for 7 days during the period between Day 8 and Day 16, and to estimate the recommended dose (RD) of C-1101.
  SyB C-1101 will be administered at a daily dose of 560 mg or 840 mg in each of the 2 cohorts for a treatment period of 1 cycle for 28 days, including 21 days for SyB C-1101 treatment followed by 7 days of follow-up.

SUMMARY:
This is a Phase 1 clinical trial to evaluate the tolerability of a combination therapy of SyB C-1101 (rigosertib sodium) and Azacytidine and to determine the recommended dose of SyB C-1101for Phase 2 trial in patients with myelodysplastic syndrome.

ELIGIBILITY:
Inclusion criteria

Patients satisfying all the following criteria will be included:

1. Histologically or cytologically diagnosed with myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemia (CMML) according to World Health Organization (WHO) Classification or French-American-British (FAB) Classification. As for patients with refractory anemia with excess of blasts in transformation (RAEB-t), however, the peripheral blood white blood cell count is ≤ 25,000 /mm3 or the state of disease was stabilized for at least 4 weeks without treatment.
2. Recognized as Intermediate-1, intermediate-2 or High according to International Prognostic Scoring System (IPSS).
3. ≥4 weeks without treatment or the effect of previous treatment (antitumor effect) is considered to be discontinued after the end of previous therapy for MDS (including using erythropoiesis-stimulating agent, ESA) or other treatment with expectation of antitumor effect.
4. Life expectancy is ≥3 months.
5. ≥20 years of age (at the time of acquiring consent).
6. Have score of 0 to 2 in Eastern Cooperative Oncology Group (ECOG) Performance Status (PS).
7. With adequate function in major organs (heart, lungs, liver, kidneys, etc.).

   * Aspartate aminotransferase (AST)(GOT): ≤3.0 times the upper boundary of the reference range at each institution
   * Alanine aminotransferase (ALT)(GPT): ≤3.0 times the upper boundary of the reference range at each institution
   * Total bilirubin: ≤1.5 times the upper boundary of the reference range at each institution
   * Serum creatinine: ≤1.5 times the upper boundary of the reference range at each institution
   * ECG: no abnormal findings requiring treatment
   * Echocardiography: no abnormal findings requiring treatment
8. Voluntarily sign the written informed consent form to participate in this study.

Exclusion criteria

Patients satisfying any of the following criteria will be excluded:

1. With anemia (haemolytic anaemia, gastrointestinal haemorrhage, etc.) caused by factors other than MDS.
2. With history or a complication of active malignant tumor (with the exception of target disease) within the past 1 year (basal cell carcinoma or squamous cell carcinoma of skin; or primary squamous cell carcinoma of the cervix or non-invasive breast cancer allows to be registered).
3. Has received administration of granulocyte colony-stimulating factor (G-CSF) within 14 days before the examination for case registration.
4. With an obvious infectious disease (including viral infections).
5. With a serious complication (liver failure, renal failure, etc.).
6. With a complication of serious heart disease (myocardial infarction, symptomatic ischemic heart disease, unstable angina, etc.). With history of arrhythmia within 2 years before registration or arrhythmia that requires treatment.
7. With a serious gastrointestinal condition (severe or significant nausea/vomiting, diarrhea, etc.)
8. Has tested positive for HBsAg or HIV antibody.
9. With serious bleeding tendencies (disseminated intravascular coagulation (DIC), internal hemorrhage, etc.).
10. With accumulation of pleural effusion/ascites that requires treatment such as paracentesis and ect.
11. With hyponatremia (serum sodium is <130 mEq/L).
12. Has undergone treatment of adrenocortical hormone (corresponding to >10 mg/24 hr of prednisolone conversion) for >2 weeks within 4 weeks before starting with administration of the study drug.
13. Has undergone treatment of another investigational product or received chemotherapy, radiotherapy or immunotherapy that was under a clinical trial stage within 3 months before the case registration .
14. Has not recovered from a surgery accompanying general anesthesia or received a surgery accompanying general anesthesia within 3 weeks before the case registration.
15. With not properly controlled hypertension (systolic pressure ≧160 mmHg or diastolic pressure ≧110 mmHg).
16. With not properly controlled epileptic seizure or with onset of epileptic seizure within 3 months before the case registration.
17. Has undergone treatment with SyB 1101 in the past.
18. With history of allergic reaction to polyethylene glycol,gelatin capsule or azacytidine.
19. Difficult to participate in the study treatment due to psychiatric disorder, social condition, ect.
20. With drug intoxication, narcotic addiction or alcohol dependency.
21. Is pregnant, nursing or possibly pregnant.
22. Is positive for pregnancy test (female patients) in the examination before the case registration.
23. Not provided consent to the following contraceptive measures. Patients should avoid sexual intercourse with sexual partners or should use the contraceptive methods as described below in the following time periods: for male patients before case registration until 6 months after the end of administration of the study drug; for female patients with menstruation before case registration until the second menstrual period is confirmed after the end of administration; for menopausal women before case registration until 2 months after the end of administration.

(1) Male patients Must always use a condom. For effective contraception, it is recommended that contraceptive methods should also be applied by the female sexual partner and patient.

(2) Female patients Must use at least 1 of the following contraceptive methods. AT the same time, the male partner must use a condom.

* Oral contraceptive (birth control pill)
* Contraceptive injection
* Contraceptive patch
* Intrauterine device (IUD)
* Tubal ligation 24. Disqualified as a subject of study treatment judged by the principal investigator or investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of dose-limiting toxicity (DLT) in patients administered with specified (level 1 or 2) dosage of SyB C-1101 in Cycle 1 and the descriptions of DLT | Up to 19 months
  Incidence rate of DLT and its binomial proportion confidence interval at the 90% level
  definition of DLT are as below: 1) Non-hematotoxicity of grade 3 or above with the exception of fever 2) fever of grade 2 or above uncontrolled by antipyretics

SECONDARY OUTCOMES:
Serious Adverse Events | Up to 19 months
Adverse Events, not including Serious Adverse Events | Up to 19 months
Change in laboratory values | Up to 19 months
Total efficacy in hematologic remission rate | Up to 19 months
  Ratio of patients scored as complete remission (CR), partial remission (PR) or marrow CR) according to the International Working Group (IWG) response criteria in myelodysplasia, 2006 (in each response criteria, responses must last at least 4 weeks):
  < CR>
  * Bone marrow: ≤5% myeloblasts with normal maturation of all cell lines.
  * Persistent dysplasia will be noted.
  * Peripheral blood:
  Hgb ≥ 11 g/dL Platelets ≥ 100 × 109/L Neutrophils ≥ 1.0 × 109/L† Blasts 0% < PR >
  All CR criteria if abnormal before treatment except:
  * Bone marrow blasts decreased by ≥ 50% over pretreatment but still > 5%
  * Cellularity and morphology not relevant <marrow CR>
  * Bone marrow: ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment
  * Peripheral blood: if hematological improvement (HI) responses, they will be noted in addition to marrow CR.
Total efficacy in hematologic improvement rate | Up to 19 months
  Ratio of patients with hematologic improvement(erythroid, platelet or neutrophil) according to the International Working Group (IWG) response criteria in myelodysplasia, 2006 (in each response criteria, responses must last at least 8 weeks):
  < Erythroid response (pretreatment, <11 g/dL) >
  1. Hgb increase by ≥1.5 g/dL.
  2. Relevant reduction of units of red blood cell (RBC) transfusions by an absolute number of at least 4 RBC transfusions/8 wk compared with the pretreatment transfusion number in the previous 8 wk. Only RBC transfusions given for a Hgb of ≤9.0 g/dL pretreatment will count in the RBC transfusion response evaluation.
  < Platelet response (pretreatment, <100 × 109/L) >
  1. Absolute increase of ≥30 × 109/L for patients starting with >20 × 109/L platelets
  2. Increase from <20 × 109/L to >20 × 109/L and by at least 100%
  < Neutrophil response (pretreatment, <1.0 × 109/L) > At least 100% increase and an absolute increase >0.5 × 109/L
Cytogenetic response rate | Up to 19 months
  Ratio of patients scored as complete cytogenetic response or partial cytogenetic response) according to the International Working Group (IWG) response criteria in myelodysplasia, 2006 (in each response criteria, responses must last at least 4 weeks):
  < Cytogenetic response > Complete: Disappearance of the chromosomal abnormality without appearance of new ones.
  Partial: At least 50% reduction of the chromosomal abnormality.
Peak plasma concentration (Cmax) | Up to 19 months
Time to maximum drug concentration time (tmax) | Up to 19 months
Area under the plasma concentration-time curve (AUC) | Up to 19 months
Elimination half-life (t1/2) | Up to 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Goto, Study Director — SymBio Pharmaceuticals
Locations (4):
- Japan (4):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Kakamigahara, Gifu
  - Research Site, Sendai, Miyagi
  - Research Site, Shinagawa, Tokyo